CLINICAL TRIAL: NCT05388188
Title: Throughput and Disposition Metrics When Using Dsuvia as a Bridging Medication to Decrease Time to Analgesia and Hospital Admissions in Patients With Sickle Cell Disease Vaso-Occlusive Crisis That Present to the Emergency Department
Brief Title: DSUVIA in Patients With SCD VOC Present in the ED
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jason Wilson (Other)
Responsible Party: Sponsor-Investigator, Jason Wilson, Principal Investigator/Medical Doctor, Tampa General Hospital
Organization: Tampa General Hospital (Other)
Other Study IDs: 20-0412
Record Dates: First submitted 2022-04-17; First posted 2022-05-24 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Sickle-Cell Disease With Crisis
Keywords: Sickle Cell Disease; SCD; SCD VOC
MeSH Terms: conditions — Vaso-Occlusive Crises; Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sickle Cell Disease Vaso-Occlusive (SCD VOC) crisis: Adult patients with known sickle cell disease present in the ED with a SCD VOC and ED provider has ordered as part of the patient's standard of care, sublingual opioid called sufentanil [Dsuvia] (a strong pain medicine that dissolves under your tongue) for the patient.
  Interventions: Drug: sublingual sufentanil
- Historical Sample: collection of retrospective data of SCD VOC patients.

INTERVENTIONS:
Drug: sublingual sufentanil — Dsuvia in patients with SCD VOC as a bridging medication.
  Other Names: Dsuvia Sublingual Product
  Groups: Sickle Cell Disease Vaso-Occlusive (SCD VOC) crisis

SUMMARY:
This is an observational study to improve the treatment of patients with Sickle Cell Disease Vaso-Occlusive Crisis by administering pain medications more quickly after the patient arrives in the emergency department. Specifically, we are using a sublingual opioid called sufentanil [Dsuvia] that has already been approved by the Food and Drug Administration (FDA) for the treatment of acute pain. It is being studied as part of this research study to find out if we can relieve the patients pain more quickly and decrease the amount of time the patient needs to spend in the hospital by avoiding a hospital admission after the patients emergency department encounter if the patients pain is adequately controlled.

DETAILED DESCRIPTION:
Patients with SCD VOC may present to the ED after oral home medications fail to relieve acute pain. Patients with SCD VOC may require parenteral analgesia for pain relief but, upon arrival to the ED these patients often undergo long wait times until receiving first parenteral medication dose. Oral opioid pain medications are not adequate as most adult patients with SCD and history of SCD VOC have already tried utilizing oral opioids out of the hospital. Intravenous access is challenging in this population with venous scarring or central ports that require sterile access. The need to establish IV access and to, eventually, provide parenteral opioids results in long delays in the time to first dose of drug (time to analgesia) in patients with SCD VOC that present to the ED. Delays in analgesia increase the likelihood of hospital admission in patients with SCD VOC that present to the ED. Patients with SCD VOC that are admitted to the hospital often have a long LOS. A bridge medication or intervention is needed for patients with SCD VOC upon entry into the ED that provides adequate and timely analgesia. In 2020, our ED began utilizing Dsuvia in patients with SCD VOC as a bridging medication. Data has not been collected to specifically examine the impact of Dsuvia use on patient throughput metrics and disposition.

Use of Dsuvia in ED patients with SCD VOC will decrease door to first analgesic time (time to analgesia). Decrease of door to first analgesic time will decrease the overall admission rate for patients with SCD VOC without decreasing patient or staff satisfaction. Use of STL Dsuvia will not lead to an increase in adverse patient safety events. Patients that receive Dsuvia early in the ED encounter may also require a lower overall amount of opioids, represented by morphine milligram equivalents (MME) than patients in a historical control group that did not receive Dsuvia. In addition, this study extends evidence for efficacy of Dsuvia in patients with acute pain but a history of opioid tolerance (unlike prior studies with Dsuvia that excluded patients with opioid tolerance). Since 2020, our ED standard of care for patients with SCD VOC is to utilize Dsuvia as early as possible in the ED course.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18
2. Known history/self-reported history of Sickle Cell Disease
3. Participant has self-described sickle cell related pain
4. Patient has attempted to utilize oral opioid pain medications in the last 24 hours

Exclusion Criteria:

1. Unable to provide informed consent to participate in the study, such as a mental condition rendering the participant unable to understand the nature, scope, and possible consequences of the study
2. Participant has a temperature of > 100.4 F
3. Participant has heart rate > 120
4. Participant has systolic blood pressure < 90
5. Clinical provider or investigator states that patient has "Acute Chest Syndrome"
6. Participant unlikely to comply with protocol as determined by Investigator
7. Clinically relevant cardiovascular, hepatic, neurological, endocrine, or other major systemic disease making implementation of the protocol or interpretation of the study results difficult or that would put the participant at risk by participating in the study
8. Persistent significant or severe infection, either acute or chronic
9. No prior oral opioid use for SCD VOC pain control
10. Participation in this study within the past 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with known sickle cell disease that present to the ED with a SCD VOC
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-03-30 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Time to Analgesia | 1 hour
  pain onset to inability to feel pain

SECONDARY OUTCOMES:
Time at Hospital | through study completion, an average of 1 week
  Length of time in the ED and/or length of stay in the hospital
Measurement of morphine milligram equivalents (MME) | 3 hours
  Total MME in patients receiving Dsuvia during ED encounter

CONTACTS AND LOCATIONS:
Overall Officials: Jason Wilson, MD, Principal Investigator — Tampa General Hospital
Locations (1):
- Tampa General Hospital, Tampa, Florida, United States